CLINICAL TRIAL: NCT04284163
Title: Learning Through Play in a University Degree: a Randomized Controlled Trial
Brief Title: Learning Through Gamification in Higher Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Daniel Ángel García, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UCAM-Gamification (PID-12/19); CE012001 (Registry Identifier: UCAM Institutional Ethics committee)
Record Dates: First submitted 2020-01-28; First posted 2020-02-25 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Motivation; Engagement, Patient
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gamification group (Experimental): Problem solving based methodology
  Interventions: Behavioral: Gamification
- Traditional teaching group (Active Comparator): Master lesson methodology
  Interventions: Behavioral: Traditional teaching

INTERVENTIONS:
Behavioral: Gamification — Teaching through gamification
  Arms: Gamification group
Behavioral: Traditional teaching — Teaching through master lesson methodology
  Arms: Traditional teaching group

SUMMARY:
"Health care legislation, management and administration" is a basic subject offered in the physical therapy university degree. The juridical features of this subject usually provokes a lack of motivation between students. Although not commonly used in university teaching, gamification could provide further affordances for improving students' engagement which provokes better assistance and learning outcomes.

DETAILED DESCRIPTION:
* 51 students of "Health legislation, management and administration" subject of the Physical Therapy University Degree of the Catholic University of Murcia will be recruited.
* Participants will be randomly assigned into two groups: control group (traditional teaching methods) and intervention group (gamification).
* Class attendance and academic results will be register for future analysis.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in the subject during academic year 19-20.
* Students included must not have taken the subject before.
* Students must be able to understand and speak the Spanish language.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Class attendance | Time-to-Event measures: from date of randomization until the end of academic period for a total of 16 week (including two holiday weeks)
  Number of days students attend class. This outcome will be registered each day by the teacher using a standardized attendance sheet template.
Total score | Outcome measures at the end of the academic period, for a total of 16 week (including two holiday weeks)
  Average score of first and second partial exams. This outcome will be obtained through qualifications in test type exam.
Partial score | Outcome measures at the end of the academic period, for a total of 16 week (including two holiday weeks)
  Score achieved in questions related to topics taught in the four intervention classes.
  This outcome will be obtained through qualifications in test type exam.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain